CLINICAL TRIAL: NCT07389057
Title: Implementation Research to Assessing the Feasibility of Combining Dihydroartemisinin Piperaquine and Primaquine for Malaria Mass Drug Administration in High Endemic Communities in the Eastern Region of Ghana
Brief Title: Assessing the Feasibility of Combining Dihydroartemisinin Piperaquine and Primaquine for Malaria Mass Drug Administration in High Endemic Communities in the Eastern Region of Ghana
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Noguchi Memorial Institute for Medical Research (Other)
Collaborators: Medical Research Center Unit The Gambia (MRCG) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NoguchiMIMR 3
Record Dates: First submitted 2026-01-12; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Malaria Asymptomatic Parasitaemia; Malaria Falciparum; Malaria Infection; Malaria Transmission
Keywords: Malaria; Mass drug administration; Ghana; Feasibility; Implementation Research
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Single Person

STUDY DESIGN:
Intervention Model Description: This is a community-randomized clinical study with a parallel design involving three arms: two intervention arms and one control arm. Eighteen communities will participate, with six communities allocated to each arm. Arm 1 will receive mass drug administration (MDA) with dihydroartemisinin-piperaquine (DHAP) alone, while Arm 2 will receive DHAP combined with a single low dose of primaquine (DHAP+PQ) to clear stage V gametocytes. Arm 3 will serve as the control with no intervention. Six rounds of MDA will be delivered bi-monthly over two years. The first round will occur 28 days after baseline, followed by 60-day intervals between subsequent rounds. If malaria prevalence falls below 5%, the second year will shift to intensive serological surveillance with targeted MDA; otherwise, MDA will continue. Treatments will be directly observed by community health workers. To assess impact, 100 participants will be randomly selected per community at baseline and follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: MDA with dihydroartemisinin-piperaquine (DHAP) alone (Active Comparator): Participants in this arm only receive DHAP. Each participants recieves one dose per day. All three doses (1 dose/day x 3days) of DHAP will be administered following NMEP guidelines. A full 3-day course of oral DHAP (40/320 mg) will be based on weight and/or age. Treatment doses will be as follow: participants weighing: (i) 5 to 10 kg (under 1 year) will received ½ tablet per day; (ii) 11 to 24 kg (1-6 years), 1 tablet per day; (iii) 24 to 50 kg (7-13 years) 1½ tablets per day and (iv) 51-70 kg (14-18 years), 2 tablets per day and ≥70 Kg (≥18 years) 3 tablets per day. All participants will be observed for 30 minutes to ensure that they retain the drug. Any participant vomiting after receiving the replacement dose will not be retreated but referred to the nearest clinic for care where necessary.
  All treated participants will be followed up on day 1, 2, 3 and 7 post-treatments to ensure to ensure adherence to treatment.
  Interventions: Drug: DHAP
- Arm 2: DHAP + Primaquine (PQ) (Active Comparator): In addition the DHAP as described in arm 1, we will add PQ. Single low dose Primaquine (0.25mg/Kg) will only be administered on day-3 to participants 10-19Kg ¼ table, 20-44kg ½ tablet, and ≥45kg 1 tablet. Under 1 years (<9Kg) children will be excluded from primaquine.
  Interventions: Drug: DHAP; Drug: Single low dose PQ
- Arm 3: Control (No Intervention): There will be no intervention in the control arm beyond the standard of care provided by health facilities in the study communities. However, at baseline and during evaluation, 100 participants will be randomly selected per community and screened for malaria parasites to determine prevalence, which will be compared with the intervention arms.

INTERVENTIONS:
Drug: DHAP — A full 3-day course of oral DHAP will be based on weight and/or age taken once daily.
  Arms: Arm 1: MDA with dihydroartemisinin-piperaquine (DHAP) alone; Arm 2: DHAP + Primaquine (PQ)
Drug: Single low dose PQ — One dose of PQ on day 3
  Arms: Arm 2: DHAP + Primaquine (PQ)

SUMMARY:
Previous malaria control studies in Ghana have shown that community-wide approaches can substantially reduce malaria infections. In a mass testing, treatment and tracking (MTTT) study, more than 75% of people in target communities were reached, leading to a 24% reduction in asymptomatic malaria after one year. However, rapid diagnostic tests (RDTs) can miss very low-level infections, meaning some infected individuals are not treated and can continue to spread malaria.

A pilot malaria mass drug administration (MDA) study using artemether-lumefantrine (AL) in the Eastern Region of Ghana showed a very large reduction (over 95%) in parasite carriage after repeated rounds of treatment. Despite this success, malaria infections later fluctuated, possibly because some parasites remained in mosquitoes and because mature gametocytes-the parasite stage responsible for transmission-are not fully eliminated by standard malaria medicines.

To better interrupt malaria transmission, this study will use MDA with dihydroartemisinin-piperaquine (DHAP) combined with a single low dose of primaquine (PQ), which targets these transmission stages. The intervention will be given to the whole community every two months (six times per year) and compared with the current standard malaria control measures.

The study will examine whether this approach reduces malaria parasite carriage, whether malaria returns after treatment stops, and whether repeated MDA affects malaria drug resistance markers in the population. This two-year implementation research will generate practical evidence to guide national malaria policy in Ghana and inform the potential use of MDA in other malaria-endemic African countries.

DETAILED DESCRIPTION:
Malaria remains the leading cause of mortality and morbidity especially among children and pregnant women in sub-Sahara Africa. In 2019 it killed 409,000 people with 67% (274,000) being under-5-years children in Africa while in 2018, Nigeria and Ghana had the highest absolute increase in malaria cases. Reducing malaria transmission by 90% by 2030 is one of the major WHO strategic goals. Recent reports reveal an upward trend of malaria prevalence in children between the age of 5 and 14 years There is renewed call to implement mass drug administration (MDA) in endemic communities which could drastically reduce the parasite level and pave the way for elimination. The Ghana National Malaria Elimination Programme (NMEP) is on track to engage malaria pre-elimination and has earmarked six districts for elimination with slide positivity rate of less than 10%. There is need to assess the impact of implementing MDA on parasitaemia prevalence in communities with holo-endemic transmission as well as resistance markers. Presently, there is paucity of data to inform the programming and implementation of MDA in Ghana. Though seasonal malaria chemoprevention is being implemented in Northern Ghana, it does not include the Southern part of the country which is holoendemic for malaria. Intermittent Preventive Treatment (IPT) of children in southern Ghana has demonstrated a parasite load reduction of over 90%.

In an ongoing mass testing, treatment and track study in Ghana, the coverage of more than 75% was achieved in target communities and reduced asymptomatic parasitaemia by 24% in one year following 4 rounds. However, in mass testing the low sensitivity of RDTs at detecting very low parasitaemia (sub-microscopic) and gametocytes leads to some cases missing treatment. Sub-microscopic parasitaemia and gametocytes are not often targeted by ACTs and can refuel transmission, hence making MDA a better option as all participants are treated. Our ongoing pilot has demonstrated that 8 rounds of MDA can reduce malaria parasite prevalence by more than 95% using AL. Could this be the case with DHAP? However, the fluctuating level of decline shows that there is a need for gametocytes to be cleared in the population for results to be sustainable. We hypothesize that implementing MDA using DHAP-alone and DHAP+PQ will reduce gametocide level and improve sustainability of reduction of parasite level.

On the other hand, there are concerns that implementing MDA in endemic communities could cause development of drug resistance due to participants not adhering to treatment. To circumvent this shortcoming, we will implement directly observed treatment (DOT). There is a need for continuous surveillance as the presence of variants of the validated markers of artemisinin resistance in the kelch 13 propeller domain of the malaria parasites has been reported in Ghana and Rwanda. Secondly, to limit continuous re-fuelling of transmission from residual parasitaemia in mosquitoes, we will conduct MDA intervention six time a year (bimonthly) as well as include a drug that target stage V gametocytes (single low dose Primaquine). The bimonthly interval is important as it reduces the potential for re-establishment of transmission when interrupted. Thirdly, we will compare the effect of using DHAP+PQ to DHAP-alone and to the standard of care in the control sites. The findings of this trial will provide data that will support policymaking. Some of the questions that need to be answered included: to what extent does MDA affect malaria asymptomatic and symptomatic parasitaemia prevalence? Does MDA affect prevalence of anaemia? Is there a possibility of a re-bound in malaria especially in under 5 children following malarias MDA? Does MDA affect the level of resistance markers in the population? What is the cost effectiveness of implementing MDA in an endemic area in Ghana? Though ongoing studies have demonstrated that MTTT is feasible and acceptable, it is not clear whether this could be the same for MDA using DHAP. The aim of this study is to assess impact of implementing MDA in endemic communities. This study will generate evidence that would inform policy on the choice of drugs and programming for the rollout of MDA in Ghana.

Serological surveillance and targeted MDA: P. falciparum is known to cause a rapid and sustained increase in variant-specific antigen (VSA) antibody levels in children. A study in The Gambia has shown that households and neighbouring compounds constitute local transmissions clusters. The acquisition of natural immunity against malaria increases with age and in Ghana anti-VSA antibodies have been reported to persist in children following infection and that some of these antigens could serve as markers of infections. A recent Gambian study has suggested that serological responses could differentiate between past and present infections as well as reflect reservoirs of infection. As malaria transmission is interrupted, the use of serological surveillance becomes inevitable in targeting asymptomatic foci of infections using MDA both at the individual and the community levels. We will use serology during surveillance for both passive and active cases. This is the first attempt to assess the impact of MDA on the population acquired immunity using serological tools for surveillance in the Pokrom sub district, Eastern Region of Ghana.

On the other hand, drug pressure presents the risk of selecting for isolates with drug resistance associated alleles and could lead to emergence of de novo resistance against artemisinins. Resistance to most partner drugs already exist, though this does not significantly affect clinical treatment outcomes with ACTs in Africa. Nonetheless, ACTs have up until this study, been mostly used for clinical management of uncomplicated malaria. The additional pressure presented by the 6 rounds of treatment requires monitoring of resistance. This is especially so in the Savannah zone of Ghana, where delayed clearance phenotype has been previously reported for some ACTs. It has been reported that widespread use of AL to treat malaria increased the frequencies of Pfmdr-1 wild alleles N86 and D126 but decreased sensitivity to lumefantrine in Uganda and Kanya it is not clear what the situation will be for DHAP. This necessitates aggressive surveillance for drug resistance markers when DHAP is use in a large scale though its efficacy in Ghana is >90% countrywide.

Objectives The primary objective of this study is to determine the effect of using DHAP-alone and DHAP+PQ for MDA on the prevalence of malaria infection in the Pokrom sub-district, Eastern Region of Ghana.

Secondary objectives

1. To determine the effect of MDA using DHAP-alone and DHAP+PQ on asymptomatic parasitaemia prevalence
2. To assess the effect of MDA on anaemia and febrile illnesses in under 15 children.
3. To genotype the plasmodium parasite in the population over time for markers of resistance.
4. To determine the challenges that impact MDA implementation.

Study site The study will be conducted in the Pokrom sub district which is one of five sub-districts in the Akwapim south district health directorate (DHD) in the Eastern region of Ghana. The Akwapim south district lies within the semi-equatorial climatic region, and experiences two rainfall seasons in a year, with an average rainfall of 125cm to 200cm. The first rainy season begins from May to June with the heaviest rainfall in June, whilst the second rainy season begins from September to October. According to the Ghana Statistical Service (GSS), the average household size in the Akwapim South district is estimated to be 4.0 whilst the average number of households per house or compound is estimated to be 1.6. The Pokrom sub district has an estimated population of 13,931 inhabitants with a malaria test positivity rate of 87%.

Stakeholder Engagement: We will organize a meeting to explain the objectives of the project and importance to all relevant stakeholders and involve them at all stages of the planning at national, regional district and community levels.

Selection and training of Community health volunteers (CHWs): 36 community health workers will be selected (2 per community) and trained on the use of RDT for malaria and treated with DHAP+PQ using the national malaria management guidelines. This training will be conducted by the National Malaria Control Programme and Ghana Health Service in collaboration with the Noguchi Memorial institute for Medical Research, University of Ghana. The CHWs will be assigned to their communities where they live and know to implement the MDA in collaboration with the research team.

All members of households in all 3 arms will be listed and a community register developed for each site.

Data collection Biological data collection: Following consent, blood will be drawn from a finger prick by trained laboratory professionals and community health workers. All participants will be tested for the presence of malaria parasites using RDTs. Additionally, 250μl of finger pricked blood will be collected on filter paper and 5 drops on a microtubule for molecular characterization of malaria parasites and genomic studies. All samples will be stored at NMIMR. For the <15-year-old subgroup study, a portable automated Hemocue photometer will be used to determine the concentration of Haemoglobin (Hb) in children. Anaemia in this study will be defined as Mild (Hb 10.0-10.9 g/dl); Moderate (Hb 7.0-9.9 g/dl); and Severe (Hb <7.0 g/dl); No anaemia (Hb >11.0 g/dl). Children with severe anaemia (Hb <7g/dl) will be referred to a health facility for follow-up. This trial will deal with all cause anaemia. Questionnaires will be used to collect data on malaria treatment, prevention, and control measures at the level of the household. Between interventions, Community health workers (CHWs) will test and treat all febrile cases.

Qualitative data collection: Data will be collected through focus group discussions (FDG), in-depth interviews, fields note, monitoring, and evaluation reports. In each community three FDGs will be conducted - one for each of the following: participants, health personnel, and CHWs. In-depth interviews will be conducted with the Heads of health facilities, district and regional health directors and selected personnel from the NMCP and GHS. FDGs and IDI will take place at prearranged venues. FGD participants will be made to sit in a semi-circle with the moderator and note taker sitting in front of them. During FGD, each participant will be given the opportunity to respond to issues posed by the moderator before progressing to another one. This will be done to ensure that all participate actively in the discussions. Participants will also be allowed and encouraged to debate and negotiate their positions to reach consensus on topical issues. Inductive probing will be used on emerging new areas. Each discussion will last within 30-60 minutes. All session will be audio taped with the consent of the participants in the local languages or English. Questionnaires will be administered to caregivers of under-15 children to assess prevalence of febrile illnesses before interventions.

Safety monitoring: In this trial we shall compare baseline to post evaluation implementation of MDA using DHAP-only and DHAP+sld-PQ; then compare DHAP group with DHAP+sld-PQ group; finally compare the difference of difference with the control group. DHAP and Primaquine are recommended for use in Ghana. Nonetheless, we shall monitor and investigate adverse events.

Adverse events reporting: Detailed information concerning adverse events will be collected and evaluated throughout the conduct of the trial. The research team will review all Adverse Event Report Forms and other interim safety data and will provide a report to the IRBs. Some participants may develop adverse reactions after taking the intervention drugs such as stomach upset, dizziness, nausea, body weakness, etc. To monitor for adverse events, participants will be followed-up by CHWs for four days (day 1, 2, 3 and 7) during and after treatment. All adverse events will be reported and referred to the health facility in the trial site. The safety of continuing the intervention will be ascertained by the participant's health care provider in collaboration with PI.

Monitoring and Evaluation: There will be monthly monitoring and evaluation visits to ensure adherence to SOPs, replenish RDT and ACT stocks, and meet with the research team, review what was done, and discuss challenges, and make recommendations. To assess the level of sub microscopic parasitaemia or gametocytes missed by RDT, microscopy will be conducted for randomly selected positive and negative participants using thin and thick film. Fifty selected confirmed microscopic samples will be verified using PCR from each community.

Data analysis

Statistical Analysis:

Baseline Comparison of Participants: Summary statistics will be produced for all variables in the study using mean (SD) and median (IQR) for continuous and proportions categorical variables. Estimation of overall malaria prevalence, the primary objective, will be done considering clustering by community; we will use random effect models to account for clustering. Additional analyses will be performed including site specific prevalence estimation as well as exploring prevalence by age group and gender. More exploratory analyses maybe performed including examining association between malaria prevalence and some potential risk factors such as age, temperature and use of nets using random effects logistic regression model.

Secondary objectives: symptomatic parasitaemia at the hospitals and symptomatic parasitaemia picked up at the community compared over time and between intervention arms using chi-square tests (or fisher exact tests) and logistic regression (or conditional logistic regression). Comparisons of anaemia in children <15 years across time and study arms will be assessed through Cochrane Armitage test of trends and using chi-square tests (or fisher exact tests) respectively. A binomial logistic regression will be used to test impact of intervention on febrile illnesses.

Qualitative data collection: Data will be collected through focus group discussions (FDG), in-depth interviews, fields note, monitoring, and evaluation reports. In each community three FDGs will be conducted - one for each of the following: participants, health personnel, and CHWs. In-depth interviews will be conducted with the Heads of health facilities, district and regional health directors and selected personnel from the NMCP and GHS

ELIGIBILITY:
Inclusion Criteria:

* must be aged 3 months and above and
* be resident in the communities for the period of the study,
* completed and signed a consent form from the parent or guardian of children below 18 years
* Completed and signed assent for 12-17 years old children.
* Completed and signed consent for those from age 18 years and above.

Exclusion Criteria:

* Pregnant women
* individual with a life-threatening illness (excluding malaria)
* less than 10Kg body weight (or less than 1 year old)
* individuals who had experienced adverse effects related to primaquine or
* known to be G6PD deficient .

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9000 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Effect of DHAP and DHAP+PQ on the prevalence of malaria infection following MDA | Time Frame: From enrolment of participants to end of treatment every two months over 24 months
  Outcomes of primary objective: asymptomatic parasitaemia will be compared over time and between intervention arms using chi-square tests (or fisher exact tests) and logistic regression (or conditional logistic regression). Adjustments for potential confounders including participant's age and use of ITN and baseline temperature will be considered. In addition, these outcomes will also be compared over time using Cochrane Armitage test of trends.

SECONDARY OUTCOMES:
Prevalence of symptomatic malaria among febrile participants attending health facilities in intervention arm compared to the control communities. | From enrolment of participants to end of treatment every two months over 24 months
  Data for symptomatic parasitaemia at the hospitals and those collected at the community will be compared over time and between intervention arms using chi-square tests (or fisher exact tests) and logistic regression (or conditional logistic regression). Adjustments for potential confounders including patient's age and use of ITN and baseline temperature will be considered. In addition, these outcomes will also be compared over time using Cochrane Armitage test of trends.
Changes prevalence of anaemia in children <15 years over time across arms | From enrolment of participants to end of treatment every two months over 24 months
  The difference in prevalence of anaemia in children <15 years in the control arm compared to the control.
  To test for anaemia in children under 15, a portable automated Hemocue photometer will be used to determine the concentration of Haemoglobin. Anaemia in this study is defined as Hb levels less than 10g/dl. Particiapnts with severe anaemia (Hb less than 7g/dl) will be referred to the Health Centre for follow up.
  Comparisons of anaemia in children <15 years across time and study arms will be assessed through Cochrane Armitage test of trends and using chi-square tests (or fisher exact tests) respectively. A binomial logistic regression will be used to test impact of intervention on febrile illnesses.
Effect of MDA on the prevalence of resistance markers. | From enrolment of participants to end of treatment every two months over 24 months
  All samples from infected individuals will be analysed for markers of anti-malarial drug resistance to explore associations between treatment intakes and presence of mutations. DNA extracts from baseline and evaluation will be analysed to determine the frequency of mutations in the Multidrug resistant protein 1 (MDR1 - N86 allele[56]), Chloroquine resistance transporter (Pfcrt - T79 Allele) and the propeller domain of Pfkelch13 (PF3D7_1343700 - C580, and C469F, K561H, R622I, A675V found in African isolates)[33, 34]. Amplicons will be sequenced, and DNA sequences will be analysed to identify specific single nucleotide polymorphisms (SNPs) related to anti-malarial resistance markers. Real time PCR analysis of the varATS gene will be used to determine the presence and quantity of P. falciparum parasites in each of the samples at the beginning and at evaluation.
Perception of the impact MDA implementation | From enrolment of participants to end of treatment every two months over 24 months
  Through qualitative research using questionnaires, focus group discussions and in-depth interviews, the population's perception of the impact MDA interventions as well as challenges affecting the process will be documented. The collected data will be transcribed and analysed thematically. A coding framework will be developed to identify key themes and patterns related to community perceptions of malaria, the effectiveness of the MDA and suggestions for improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Ndong Ignatius Cheng, PhD, Principal Investigator — Noguchi Memorial institute for Medical Research, College of Health Sciences, University of Ghana
Locations (1):
- Pokrom sub district, Accra, Eastern Region, Ghana

IPD SHARING:
Plan to Share IPD: No
Participant data collected under this project is confidential. It is an IRD requirement not to share participant data.